CLINICAL TRIAL: NCT02809651
Title: A Prospective Study to Determine Confounding Factors in the Detection of Intracranial Hemorrhage With the Infrascanner
Brief Title: Confounding Factors in the Detection of Intracranial Hemorrhage With the Infrascanner
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Pascal Vanelderen, Prof. Dr., Ziekenhuis Oost-Limburg
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 16/015U
Record Dates: First submitted 2016-06-18; First posted 2016-06-22 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Ischemic Stroke; Brain Tumor; Brain Surgery; Intracranial Hemorrhage; Headache; Head Trauma
Keywords: Infrascanner; Intracranial hemorrhage
MeSH Terms: conditions — Ischemic Stroke; Brain Neoplasms; Intracranial Hemorrhages; Headache; Craniocerebral Trauma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Ischemic stroke (Experimental): patients suffering from ischemic stroke diagnosed by clinical examination and CT-scan
  Interventions: Device: Infrascanner
- Brain tumor (Experimental): patients diagnosed with a brain tumor diagnosed by clinical examination and CT-scan or MRI
  Interventions: Device: Infrascanner
- Brain surgery (Experimental): patients that have undergone brain surgery
  Interventions: Device: Infrascanner
- Intracranial hemorrhage (Active Comparator): patients with intracranial hemorrhage diagnosed by clinical examination and CT-scan
  Interventions: Device: Infrascanner
- Headache (Experimental): patients with headache complaints and a normal CT-scan of the brain
  Interventions: Device: Infrascanner
- Headtrauma (Experimental): patients with head trauma and a normal CT-scan of the brain
  Interventions: Device: Infrascanner

INTERVENTIONS:
Device: Infrascanner — bilateral measurement cerebral blood flow with near infrared spectroscopy using the Infrascanner on the frontal, temporal, parietal and occipital region of the head.

SUMMARY:
The investigators prospectively want to use the Infrascanner in patients with ischemic stroke, patients with brain surgery, patients with brain tumors, patients with intracranial hemorrhage and patients with a normal CT scan of the brain as part of a diagnostic work-up after head trauma or headache to determine to positive and negative predictive value of the Infrascanner in these different settings.

DETAILED DESCRIPTION:
Infrascanner is a portable device initially designed to detect intracranial hemorrhage in battlefield traumas. Infrascanner uses near infrared spectroscopy to measure cerebral blood flow non-invasively. This is achieved by putting the device against the scalp in 4 different areas (frontal, temporal, parietal, occipital) on the left and right side and by comparing both sides.This allows for the detection of intracranial hemorrhages with a volume upwards of 3.5ml and to a depth of 2.5cm. However, little is known about the influence of other intracranial conditions that could confound the measurements of the Infrascanner (e.g. ischemic stroke, brain surgery, brain tumors,...).

Therefore, the investigators prospectively want to use the Infrascanner in patients with ischemic stroke, patients with brain surgery, patients with brain tumors, patients with intracranial hemorrhage and patients with a normal CT scan of the brain as part of a diagnostic work-up after head trauma or headache to determine the positive and negative predictive value of the Infrascanner in these different settings.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ischemic stroke diagnosed by clinical examination and CT-scan
* Patients with a brain tumor diagnosed by clinical examination and CT-scan or MRI
* Patients with an intracranial hemorrhage diagnosed by clinical examination and CT-scan
* Patients that have undergone brain surgery
* Patients with a normal CT-scan of the brain after head trauma
* Patients with headache complaints and a normal CT-scan of the brain as part of their diagnostic work-up

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2016-08; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Presence of intracranial hemorrhage as indicated by the Infrascanner compared to the result of the CT-scan (gold standard) | 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Vanelderen, MD, PhD, Principal Investigator — member of Staff
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No